CLINICAL TRIAL: NCT00811499
Title: A Study of ARRY-371797 in Patients With Active Ankylosing Spondylitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARRAY-797-201; C4411006 (Other: Pfizer)
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — ARRY-371797

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARRY-371797 (Schedule 1) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- ARRY-371797 (Schedule 2) (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral; Drug: Placebo; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — multiple dose, single schedule
  Arms: ARRY-371797 (Schedule 1); ARRY-371797 (Schedule 2)
Drug: Placebo; oral — matching placebo
  Arms: Placebo
Drug: Placebo; oral — multiple dose, single schedule
  Arms: ARRY-371797 (Schedule 2)

SUMMARY:
This is a Phase 2 study, involving a 12-week treatment period, designed to evaluate the effectiveness of investigational study drug ARRY-371797 (versus placebo) in treating ankylosing spondylitis, and to further evaluate the drug's safety. Approximately 130 patients from the US, Canada, Poland and Hungary will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of ankylosing spondylitis according to the Modified New York Criteria (1984).
* Inadequate response to at least 2 weeks of continuous treatment with NSAIDs, or unable to receive ≥ 2 full weeks of continuous treatment with NSAIDs because of intolerance.
* If previously treated with a biological agent, patient must not have failed due to lack of efficacy, and must have completed an appropriate washout period prior to first dose of study drug.
* Patients may continue on specified stable background therapies for ankylosing spondylitis (doses should be stable for at least 4 weeks prior to the first dose of study drug).
* Additional criteria exist.

Key Exclusion Criteria:

* Diagnosis of any other active or uncontrolled inflammatory or non-inflammatory articular disease that may interfere with disease activity assessments.
* Previously treated with intravenous immunoglobulins within 6 months prior to first dose of study drug.
* Patients requiring prohibited concomitant medications including moderate or strong CYP3A inhibitors, CYP3A inducers and Biologic Response Modifiers (BRMs) while on study.
* Trauma or other major surgeries within 8 weeks prior to first dose of study drug.
* Specific abnormal laboratory values or electrocardiogram abnormalities.
* Known positive serology for human immunodeficiency virus (HIV), hepatitis C, and/or hepatitis B.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12-16 (Actual); Primary Completion 2009-09-29 (Actual); Study Completion 2009-09-29 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug (versus placebo) in terms of Assessments in Ankylosing Spondylitis 20% Working Group response criterion (ASAS 20). | 12 weeks
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | 12 weeks

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) of the study drug and a metabolite in terms of plasma concentrations. | 12 weeks
Explore potential biomarkers for pharmacodynamics (PD). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Westroads Medical Group, Omaha, Nebraska
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Low Country Rheumatology, Charleston, South Carolina
  - Arthritis Northwest, Spokane, Washington
- Canada (5):
  - Rheumatology Research Associates Group, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Credit Valley Rheumatology, Mississauga, Ontario
  - Center de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests